CLINICAL TRIAL: NCT00949143
Title: Effects of Axle Positions on Wheelchair Skills in Manual Wheelchair Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Dr. R. Lee Kirby, Capital District Health Authority
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: CDHA-RS-2009-182
Record Dates: First submitted 2009-07-28; First posted 2009-07-30 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Physical Disability
Keywords: wheelchair user

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- forward position (Experimental)
  Interventions: Other: forward axle position
- rear position (Experimental)
  Interventions: Other: rear axle position

INTERVENTIONS:
Other: rear axle position — Wheelchair axle position located as far towards the rear of the wheelchair as possible.
  Arms: rear position
Other: forward axle position — Wheelchair will have the axle at least 5cm farther forward than the most rear axle position.
  Arms: forward position

SUMMARY:
The aim of this study is to investigate the effects of altering the wheelchair set-up on mobility and safety by changing the rear-axle position on a manual wheelchair.

ELIGIBILITY:
Inclusion Criteria:

* manual wheelchair users
* minimum of 17 years of age
* at least one week experience in a manual wheelchair, for at least an hour a day
* alert
* able to answer questions
* able to fit in the testing wheelchairs
* permission to participate from the attending physician

Exclusion Criteria:

* significant visual impairments
* unstable medical conditions (e.g., angina)
* emotional/psychological problems that may make testing unpleasant

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Wheelchair skills test | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Lee Kirby, MD FRCPC, Principal Investigator — CDHA
Locations (1):
- Nova Scotia Rehabilitation Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- See also: Related Info — http://www.wheelchairskillsprogram.ca